CLINICAL TRIAL: NCT02033915
Title: The Effectiveness of Interactive Discussion Group Intervention to Improve Nurses' Abilities of Risk Identification and Assessment on People With Suicide Attempt or Self-harm Behavior
Brief Title: The Effectiveness of Interactive Discussion Group Intervention About Suicide Risk Identification and Assessment for Clinical Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 201107036RB
Record Dates: First submitted 2011-10-07; First posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Suicide Risk Assessment
Keywords: Suicide risk assessment; interactive discussion group; suicide attempt; self-harm; randomized control study; identifying high risk group for suicide
MeSH Terms: conditions — Suicide, Attempted; Self-Injurious Behavior

ARMS (1):
- Interactive Discussion Group (Experimental): The interactive discussion groups were held for six times (8-10 persons for each group). During the 50-60 minutes' discussion, the facilitators guided the participants to discuss a case vignette, focusing on the key issues of hospital suicide prevention, and to enhance their abilities of suicide risk identification and evaluation. Two research team members who served as facilitators led the group in a standardized manner.
  Interventions: Other: Interactive discussion group

INTERVENTIONS:
Other: Interactive discussion group — The investigators adopt the group intervention that provide interactive discussions regarding the assessment of suicide risk among inpatients in a general hospital.

SUMMARY:
Suicide attempters or people with self-harm have a high percentage in seeking medical services before and after their suicidal or self-harm behaviour compared to general population. Studies revealed that apart from psychiatric services, they were more likely to seek help from doctors of various units (e.g. emergency departments, general medicine, medical-surgical units) across different healthcare systems (i.e. hospitals or district clinics). Besides, suicide event was possibly heard on in-patients of psychiatric or non-psychiatric units. People with self-harm experienced poor communication with healthcare personnel, and they perceived staff's lacking knowledge about suicide as serious problems. In Taiwan it was also found that emergency nurses and general practitioners were in need of improving negative attitudes and enhancing knowledge towards suicidal behaviour. From the point that nurses are the healthcare personnel that spend the most time with in-patients compared to others in the hospital, suicide risk assessment training may enhance nurses' attitudes and ability of risk awareness and assessment towards people with self-harm, which may in turn significantly increase the identification rate of the high risk group for suicide. Currently there is a lack of suicide training program as a reference for nursing education in Taiwan. The study therefore aims to strengthen suicide risk assessment ability among clinical nurses through interactive discussion groups. Using quasi-experimental design with randomized cluster sampling strategy, a case vignettes will be used for suicide risk assessment together with other measurements regarding suicide knowledge and attitudes for both experiment and control groups before and after the training course.

DETAILED DESCRIPTION:
Title:

The effectiveness of interactive discussion group intervention to improve nurses' abilities of risk identification and assessment on people with suicide attempt or self-harm behavior

A.Background

Suicide has become an important issue in the public health and medical-related field in the past decade and has also aroused the attention of government in Taiwan. It has been one of the top ten cause of death since 1997 . The high percentage of people who act on suicide idea in different age groups pose great challenge to healthcare personnel. Clinical workers are first-line gatekeepers of patient health and safety. They are supposed to be willing to care for people with suicide risk and can be equipped with the ability to identify patients with suicide risk. However, the negative attitudes of medical workers towards people who have suicide attempt and self-harm behavior may affect the patients' intention to seek professional help and the nurses' quality of care for these people . At present, the investigators have limited nursing curriculum related to the concept of and guidance for suicide prevention and limited resources that guide nurses to do suicide risk assessment. Few information about suicide process and suicide risks are available for nurses , which may result in their inability to provide proper care for this group of people. If the investigators can improve the ability of suicide risk identification of the nurses, the investigators may promote nurses' confidence and change their attitudes in caring for such patients. Also, nurses can learn how to empathize suicidal patients, intervene at early stage of patients' hospitalization, and potentially build good nurse-patient relationship with patients under high risk for suicide. Furthermore, the investigators can refer patients to receive appropriate therapy and to provide adequate support to reduce their suicide attempts. The investigators addressed the background and importance of this study in the following sub-sections:

The importance of suicide prevention throughout the process of nursing education and clinical training

People with deliberate self harm behavior are the high risk group for suicide, and the prevalence of self-harm behavior is 10-30 times to suicide . Identification and assessment of suicide risk is the main target of suicide prevention. However, there are only few opportunities for nurses to acquire knowledge about suicide prevention in the process of nursing education and training. For instance, in a Nursing Department of Medical college in Northern Taiwan, there is only one class talking about related issue of suicide prevention among all the Psychiatric Nursing lectures. In general, student nurses think they are unfamiliar with this issue and unable to assess the patients' suicide risk. Clinical nurses who have more chance to care for suicide high risk group, such as those in the Emergency Department (ED) and psychiatric ward, may still have negative attitudes toward self-harm behavior. Nurses regarded suicidal behavior as selfish, wasting of social or medical expenses, or not worthy of showing sympathy. Moreover, they may think self-harm behavior as a kind of controlling behavior, calling for attention, and difficult in caring or building therapeutic relationship. These negative thinking and emotions are both less likely to promote caring quality to patients with self-harm. It was found that psychiatric nurses tended to use verbal communication, to inform doctors about patients' suicide risk, or to give close observations to prevent self-harm act or to offer a safe environment in the psychiatric ward. But there is a lack of concept of early prevention among clinical nurses, irrespective those working in the psychiatric or medical-surgical wards. Patients who suffer from chronic illness or in terminal stage of disease in medical wards might have more suicide ideations. It might be helpful to promote the ability of suicide identification and assessment among nurses to give better caring quality for the suicide high risk population. Moreover, nurses in the ED are easily encountered with the high risk (i.e. people who had suicide attempt or self-harm behavior before). There is still few research focusing on the ability of suicide risk evaluation of nurses in the ED. It was suggested that training courses can change the negative attitude of suicide for nurses who work in the ED, promote their ability of suicide risk assessment, and enhance their confidence in facing these patients.

The policy of suicide prevention and gatekeeper program are forming currently by the health organization in Taiwan. Not only are the public playing the role of gatekeepers to indentify suicide risk, clinical nurses should also know how to assess suicide risk. So far the investigators have few courses about suicide risk assessment, and the investigators need further research to develop a complete content of suicide evaluation, which can be used in clinical training and nursing education. The investigators can provide a learning environment based on interactive group, and this can help improve critical thinking and problem solving skills. Also, using case vignette to design the discussion course (case-based curriculum) can help the learners understand integrated knowledge content based on clinical situation; its advantages include to promote the motivation of active learning, to strengthen the analysis skills, to enhance decision making ability, or to cultivate learners o how to correctly evaluate the effects on patients from social culture perspectives. At the present, nursing education in Taiwan is focusing on critical thinging, problem-solving, and decision making, and the use of group discussion can help reach the above teaching goals.

The importance of patient safety in hospitals

It is important to keep patient safety in the medical environment, and it is also necessary to provide quality of care. However, the issues of suicide and self-harm behavior have been neglected in hospitals, and the investigators are lacking of effective preventive interventions and policy. There are many topics related to patient safety in medical environments, including mistakes happened during the process of giving medicine, falling, environment safety. However, suicide behavior among inpatients has been posing the greatest challenge to medical personnel. According to the Taiwan Patient-Safety Reporting System (Taiwan Joint Commission on Hospital Accreditation, 2009), there were 1,613 accident events of hospitalized patients in 2008. General wards are the mainly location of events, in the categories of events, 12.0% is self-harm behavior. Although there are only 43 events of suicide attempt, its consequence are the most serious compared to other patient safety issues. Researches in the 1960s in western countries indicated that the death rate of suicide among hospitalized patients are 0.06~5.66 per thousand. Even suicide is a rare topic, the investigators cannot ignore its severity. To prevent suicide events, psychiatric ward and general ward should put emphasis on the prevention, the education training and communications between patients and nurses (Taiwan Joint Commission on Hospital Accreditation, 2009). For general medical workers, they might underestimate the formation and the effects of suicide or self-harm behavior. The investigators may reach the goal of suicide prevention and treating for self-harm behavior appropriately if clinical nurses can identify the high risk group of suicide effectively and follow the steps suggested in the gatekeeper program.

The importance of suicide risk assessment

There is a remarkable percentage seeking for medical help among patients who harmed themselves before committing suicide. These patients not only appeared in psychiatric department, but also seek medical help in different medical settings. According to a systemic literature review, people of self-harm behavior think they do not have good communication with medical workers, and most medical workers do not have idea about what self-harm behavior is either. This is a common problem in the medical system across different departments. The investigators also understand that negative attitude or knowledge do actually exist in the nurses of Emergency Department and doctors. Tzeng & Lipson (2005) suggested that medical workers need to know the reasons of suicide or self-harm behavior and the kind of interventions that may be helpful. Cognition and attitude training like this is not usual in nursing education, but nurses, among the medical group, have relatively more time to stay with patients. So strengthen the training of suicide evaluation and identification can help us to know the potential group of high risk, and also provide social support and medical connections to reduce the formation rate of suicide and self-harm behavior.

The reasons why the investigators need to identify and assess suicide risk

To identify and evaluate the suicide risk is the first step in suicide prevention. Evaluations for factors of suicide risk (such as major depression and high risk group of suicide)is not often performed in clinical care, expect for the psychiatric care settings. However, the process of help seeking behavior could happened in the following ways such as self-disclosure of suicide idea and risk factors, or transferred by nurses in any department and start to accept further treatment. In this process, help and social support from family or friends can strengthen the intention to seek for help. Therefore, to identify the case with potential risk is the key point to start suicide prevention. Although the investigators don't have any research talking about suicide prevention policy in hospital now in the world, the awareness and identification for group with high risk, risk assessment and transfer are strongly recommended by many Western countries. Nurses can play the role of gatekeeper of suicide prevention, and identify the suicide or self-harm behavior before it occurs and transfer to the right association for further caring instead of providing assessment and protective instructions after the event.

Based on the backgrounds, this research focuses on the ability of suicide risk identification and evaluation of clinical nurses in a teaching hospital of Northern Taiwan. And the investigators do evaluate the impact of interactive discussion group which promote the identification ability for nurses. The investigators expect to find out patients with high risk of suicide and provide appropriate interventions by improving the sensitivity of first line clinical professionals.

B. Aims of the study

* To improve the ability of suicide risk identification and assessment on hospitalized patients for clinical nurses
* To understand the impact of using the interactive discussion group to promote the ability on suicide risk identification and evaluation for clinical nurses
* To provide evidence-based nursing education as a basis to practice the interactive discussion group to promote nurses' ability on suicide risk identification and evaluation

C. Methods

The study is a randomized controlled trial. The sample will be consisted of 120 people, with half of them allocated to the intervention group and another half allocated to the control group. Therefore, the sample will be distributed into experimental group and control group equally and randomly. After receiving approval from the Ethical Review Committee, the investigators will start recruiting people to attend the intervention, "interactive discussion group" (IDG), the investigators aim to discuss the concept of suicide risk identification and evaluation as well as investigate the impact of such an intervention. The investigators have developed a standardized teaching program (the IDG and suicide gatekeeper course for nurses) as our intervention. Moreover, before starting the intervention, the investigators will have three focus groups in the pilot study in order to recruit clinical nurses' perspectives on the issue of the study and their opinions of the study tool. Depends on their opinions, the investigators will revise the teaching materials and assessment tools, and evaluate the feasibility of putting the IDG into practice. Next, the experimental group will take one suicide gatekeeper course and the IDG discussion twice, and the control group takes one suicide gatekeeper course. The investigators will do the baseline measurement and outcome measurement to evaluate the effects of intervention. The research methods and rationale are described in details below.

The rationale of adopting the intervention of "interactive discussion group" (IDG)

Education training for nurses currently includes classroom teaching through speeches, film/website teaching, group discussion and practice, and classroom teaching is most popular one in nowadays. Materials the investigators use to teach suicide assessment such as interactive website which provided by Taiwan Nurses Association and books are also available for nurses for self-learning. Concerning the importance of discussion and evaluation of suicide risk, and the realization of suicide risk based on a case vignette, also the interactive learning between trainees and facilitators, the investigators choose using interactive discussion group as our teaching policy, and via the randomized controlled trial the investigators can evaluate the effect or research interventions.

Standardized procedure of the interactive discussion group

Researchers will take the interactive discussion group class for six times (8-10 persons every time). During the 50-60 minutes, the facilitators will guide the trainees to understand the case vignette and focus on the key issues to discuss, to improve the ability of suicide risk identification and evaluation. Two research team workers are responsible for the facilitators, and they are both experienced in suicide prevention and clinical works. The two facilitators will guide the group in a comprehensive way and standardized maneuver. The topic of discussion is focus on a suicide case, a 47-year-old man, who is now in hospitalization of medical ward. In the content the investigators can find out there are many messages and signs of major depression and suicide behavior. Through the discussion, the investigators guide nurses to realize the suicide-related factors, and teach them to identify/evaluate the suicide risk. 10 minutes before the group, the investigators ask the trainees to read the case and answer the questions. In the next 30 minutes, the investigators start problem discussion and use three simple, convenient tools: PHQ2, simplified health scale, SAD PERSONS, to do the teaching of identification and evaluation of suicide risk. In the last 10-15 minutes, the investigators go into a conclusion, do point review and get feedback from trainees.

The Research team uses the standardized material course which is authorized by the Health Department of Taiwan-"The Gatekeeper Training Program" to do our interventions. Facilitators are trained to use the same material and ways to teach the experimental group and control group in consistency. In this part, the investigators do not discuss the suicide case vignette, so the investigators can divide this from the group which trained by interactive discussion and therefore the investigators can evaluated the effect of using discussion group in our training.

Research Tools

1. The baseline measurement 1-1 Information Assessment of basic demographic variable such as age, sex, marriage, duration of practicing in nursing, nursing levels, working experience of psychiatric wards, caring experience of person they know (friends, colleague or neighbors) or patient who committed suicide or self-harm behavior before, do they accept any training related to suicide prevention in the past year.

   1-2 Suicide Case vignettes and risk assessment question Research team designed a case discussion depends on clinical experiences and suicide cases they had cared before. The investigators drafted some important questions to evaluate the ability of suicide risk identification and evaluation of research samples (Nurses). 8 student nurses of university went through this case discussion, and the investigators got a good result of this pilot test. Student nurses all agreed the interactive discussion with teacher and problem-based teaching can help them to grab the point of suicide prevention and arouse their learning interest.

   1-3 Assessment of the cognition and attitude to suicide behavior This scale is used in the survey by Health Department of Taiwan which to understand the attitude and opinion toward suicide and Psychiatric disease of randomized sample size in the population of Taiwan. And the validity of this tool was already proved.
2. Assessment tools in the Interactive Discussion Group 2-1 Case vignette is the point in our interactive discussion group, please read the details in <Methods>.

2-2 PHQ PHQ was originally used to evaluate the health situation of general public in community, and PHQ-9, a part of this scale, which used to evaluate the tendency of Major Depression. And the content of PHQ-9 is correlated to the 9 diagnosis items with DSM IV. Scholars modified a new vision of PHQ-2, and the reliability and validity is good on the public of Taiwan (Sensitivity: 88.0%, Specificity: 81.9%) (Lu et al., 2010). Therefore the investigators use the scale to train nurses to screen if there is possibility of Major Depression in patients. The two questions are related to the symptoms of "depressed mood" and "lost of interest".

2-3 Simplified Health Measurement Scale This scale is developed to test the general mental health of the public, including five question as "do you feel nervous and anxious", "easily to feel worrisome and angry", "feeling depressed and sad", "feeling of low self-esteem" and "bad sleeping quality". Also, the investigators ask extra question as "do you have any suicide idea". This reliability and validity was proved by Li et al.,(2003), and it's a simple, convenient scale to screen out the potential depression tendency and suicide risk. The goal the investigators use this scale in the research is to improve the recognitions of nurses on Major Depression.

2-4 SAD PERSONS-check list of suicide risk This checklist was originally designed to screen if a patient needs to be hospitalized by the Emergency Department staffs based on a 10-item suicide risk screening sheet.

S - Sex: male A - Age( <19 or >45) D - Depressive symptoms P - Previous suicide attempt/psychiatric care E- Excessive ethanol/drug use R- Rational thinking loss, sever psychiatric symptoms as delusion, hallucination S - Separated/ divorce/drug use/widowed O - Organized or serious attempt, who had severe and objective self-harm behavior before like carbon monoxide poisoning, overdose medicine taking and need to be hospitalized…etc.

N - No social support, lack of family, friends, work and religion support S - Stated future intent, clear plan including time, methods and location

Each item is scored one point, with two points weighing for items that are underlined. Kripalani et al., (2010) suggested people who get five points or higher need to be hospitalized and accept further therapy. The validation of the Chinese version of the scale has been performed by a group of psychiatric researchers in Taiwan and is under drafting.

Data collection procedure

1. The target population and study sample The target population (i.e. clinical nurses) for the study is defined to be from a variety of ward such as Hematology, Oncology, Stroke and Rehabilitation where potential cases with high suicide risk may be identified. The investigators hypothesise that nurses who work in these wards should understand more about the concept of suicide prevention and suicide risk assessment. Therefore the study will include all clinical nurses in these wards as the target population. The sample size is calculated based on the suggestion in the literature, and the investigators set the significant level data, α = 0.05, power = 0.80. Then the investigators divide all study subjects into experimental group and control group randomly, and use different interventions to examine the effect of research.
2. Pilot study

   The investigators design focus group courses (three times) for clinical nurses to understand their opinions and needs about the teaching materials of suicide risk identification and assessment. Also, the investigators examine the possibility of adding the interactive discussion group which suggested by group discussion. The investigators choose 6-8 nurses each time out of the study samples randomly and excluded who had already joined the focus group before. Location of the focus group is on the independent discussion room in hospital. Meanwhile, nurses who joined focus group will also be excluded in the later study samples (neither the experimental group nor the control group).
3. The baseline measurement

   The experimental group and control group will both be administered the baseline measurement including the ability of suicide risk identification, attitude and recognition toward suicide behavior, and the ability of suicide risk assessment (the investigators use a case vignette and the SAD PERSONS check list). The goal of baseline measurement is to evaluate the difference of demographic characteristics and perceptions and attitude toward suicidal behaviour between the two research groups before the intervention.
4. The outcome measure

The investigators will use the score of SAD PERSONS-check list as the outcome measure in assessing the effect of our intervention. The reason of using this check list is because it is a simple and convenient tool to screen suicide risk in clinical settings, and researches have proofed its reliability and validity.

Statistical analysis

All statistic analysis of this research are based on the Intent-to-treat method, which follow up participants who cannot finish the whole study process (i.e. drop out from the study). The investigators still ask them to do the outcome measurement. All the data will be count into the original groups to do further analysis in order to get a conservative conclusion. Researchers will key-in the data the investigators will use SPSS 16.0 to do the statistical analysis. The significant level will be set at 0.05. Main variables and methods for analysis are listed below:

Independent variables

1. Demographic information: Basic demographic variable such as age, sex, marriage status, nursing practice years (continuous variable); categorical variables such as nursing levels recognized in the study hospital, working experience in psychiatric related field, caring experience of suicidal persons of their acquaintances (friends, colleague or neighbors) or patient who committed suicide or self-harm behavior before, training experiences related to suicide prevention in the past year.
2. Variables in the baseline measurement: Attitude and cognition toward suicide (continuous variable), the ability of suicide risk identification and assessment (category variables), and SAD PERSONS-the check list of suicide risk (continuous variable).

Outcome variables The ability to identify and evaluate the suicide risk, SAD PERSONS-the check list of suicide risk (continuous variable), and case analysis 1(category variable)

Baseline comparison To make sure there is no difference at first among participants in this research, the investigators will compare the characteristics and basic ability of suicide risk. Independent t-test is used to deal with continuous variables, and Chi-square test is used for category variables. However, whether there is significant difference or not, the investigators will further analyze their suicide identification and assessment ability in multivariate analysis.

Further analysis The investigators will compare the change in scores of the outcome, the scale of "SAD PERSONS", as the continuous variables before and after the interventions. The investigators will also analyze the frequency and associations of the items in baseline measurement including the participants' working site, age, sex, education, duration of nursing practice, trainings of suicide risk assessment, caring experience of suicide or self-harm cases.

D. Predictable Difficulties and Solutions

1. Attendance and Participation of the interactive discussion group in Nurses According to the different shifts of clinical nurses, before the investigators arrange the schedule of interactive discussion group, the investigators will completely communicate with chief manager of different department and get the support of hospital administration to make sure that the investigators have an appropriate time for every member in the group. Also, researcher will remind of every member one by one to elevate the attendance and participation. Furthermore, all the time nurses spend on this training will be count into the in-service education time to arouse enforce the motivation. Besides, researcher will provide the research fee to every participant to promote the participation interest.
2. Missing data in the questionnaire To prevent the missing data, the researchers will join every discussion activity to examine if there is any problem for nurses to fill out the questionnaire, and keyin the data individually to ensure its correctness. Moreover, the research assistant will key in the data twice under surveilance of the principle investigator during the whole procedure.

ELIGIBILITY:
Inclusion Criteria:

* nurses who work in a variety of wards such as Hematology, Oncology, Stroke and Rehabilitation where potential cases with high suicide risk may be identified.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Correctness rate and the scores of the nurses to identify the risk factors of a case vignette using an assessment tool, the SAD PERSONS Scale. | 12 months
  The study aims to strengthen suicide risk assessment ability among clinical nurses through training group discussions. In the group sessions the nurses will be facilitated to discuss the suicide risk factors of a case vignette and use an assessment tool, the SAD PERSONS Scale, to learn those factors. The primary outcome measures will be the correctness rate and scores the nurses ascertained in suicide risk assessment of both groups. We hypothesise that the experimental group will have higher correctness rate after the study intervention.

SECONDARY OUTCOMES:
(untitled outcome) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Yi Wu, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- Chia-Yi Wu, Taipei, Taiwan